CLINICAL TRIAL: NCT05345314
Title: Endoscopic Grading of Gastric Intestinal Metaplasia: a Validation Study in Korea
Brief Title: Endoscopic Grading of Intestinal Metaplasia
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-EGD-2022
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Narrow-band Imaging; Magnifying Endoscopy; Gastric Intestinal Metaplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen would be obtained for pathological analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Narrow-band imaging endoscopy — During endoscopy, gastric mucosal patterns would be examined by magnifying narrow-band imaging.

SUMMARY:
Long-term Helicobacter pylori infection causes premalignant gastric conditions, such as atrophic gastritis and intestinal metaplasia. Image-enhanced endoscopy techniques such as narrow-band imaging (NBI) and magnifying endoscopy improve the diagnosis of gastric intestinal metaplasia (GIM). However, there are no comparative data on the utility of NBI and magnifying endoscopy for diagnosing GIM.

DETAILED DESCRIPTION:
This study aims to evaluate the diagnostic performance of NBI and magnifying endoscopy for GIM in a country with high risk of gastric premalignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* Pathological analysis can be performed for analysis of gastric atrophy and intestinal metaplasia

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2-receptor antagonists, or antibiotics
* History of H. pylori eradication
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All of the patients underwent gastroscopy for peptic ulcer, gastric cancer screening in a single academic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Gastric intestinal metaplasia | 4 weeks
  Gastric intestinal metaplasia would be assessed using pathological examination.

SECONDARY OUTCOMES:
Degree of chronic gastritis | 4 weeks
  Gastric atrophy would be evaluated on the basis of histopathological examination (updated Sydney system).

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No